CLINICAL TRIAL: NCT03321682
Title: Cardiopulmonary Capacity and Quality of Life in Patients With Chronic Heart Failure Submitted to Functional Training - a Randomized Clinical Trial
Brief Title: Cardiopulmonary Capacity and Quality of Life in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69314017.8.0000.5327
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Cardiopulmonary Capacity; Quality of Life; Functional Capacity; Functional Training
MeSH Terms: conditions — Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Training (Experimental): Patients in the functional training group, in addition to maintaining their usual care, will perform functional training including exercises for core strength, power training, knee dominance, hip dominance, horizontal pressure, vertical pressure, horizontal pull and vertical pull, using unstable surfaces.
  Interventions: Other: Functional Training
- Strength Training (Active Comparator): These group, in addition to maintaining their usual care, will perform the exercise protocol as recommended by the American Heart Association.
  Interventions: Other: Strength Training

INTERVENTIONS:
Other: Functional Training — Exercises performed in circuit, using weights, elastic bands, suspension tapes, cones and on unstable surfaces.
  Arms: Functional Training
Other: Strength Training — Exercises carried out using weights and involving the main muscle groups.
  Arms: Strength Training

SUMMARY:
Heart Failure is a progressive disorder that begins after an insult to the heart muscle resulting in the loss of functional cardiomyocytes, or even compromising the ability of the myocardium to contract and/or relax normally. A common finding in heart failure is exercise intolerance that generates a vicious cycle, in which the individual starts to limit his activities even further due to progressive fatigue. Studies demonstrate that regular physical exercise can increase the aerobic capacity of these individuals, delay the anaerobic threshold, and reestablish the sympathovagal balance. Paradoxically, many of these patients assume an even more sedentary lifestyle, which leads to a greater physical limitation and the progression of symptoms. Patients with heart failure present a 30% reduction in their ability to perform their daily life activities when compared to healthy individuals, and this has also been attributed to reduced muscle mass, as well as lower aerobic capacity. In this sense, strength training increases the torque and muscular endurance, capacity and functional independence, as well as the quality of life, reducing the morbidity of individuals with and without cardiovascular disease, with a lower overload to the cardiorespiratory system. It is known, however, that daily life activities require a combination of resistance and muscle strength. Aerobic training does not improve muscle strength, just as traditional strength training does not ideally represent the movements performed during daily life activities, since it does not include exercises on unstable surfaces and exercises on different axes. Functional training emerges as a simple and low cost alternative for the treatment of patients with heart failure. This method consists of integrated movements of the body, in several axes, involving joint acceleration and deceleration, stabilization, strength and neuromuscular efficiency. It aims to improve the functional capacity of the individual using exercises that relate to their specific physical activity, transferring their gains effectively to their daily lives. The aim of the present study is to evaluate the effects of functional training on cardiopulmonary capacity and quality of life in patients with heart failure, comparing it to strength training.

DETAILED DESCRIPTION:
Individuals with cardiac heart failure, in functional class II and III (according to the New York Heart Association), residents of the metropolitan region of Porto Alegre, of both genders and aged ≥ 18 years, will be recruited from the Outpatient Clinical of Heart Failure of the Hospital de Clínicas of Porto Alegre, RS/ Brazil. At the end of the initial evaluations of each participant, they will be randomly allocated in one of two groups: functional training group (FTG) and strength training group (STG). After the consent of the participants, the author of the research will start collecting the data, by completing an anamnesis form. The following evaluations will be performed before the start of the study and immediately after the end of the research, by prior appointment: cardiopulmonary capacity, quality of life, functionality, palmar grip strength, maximum inspiratory pressure, endothelial function and lean body mass. Both groups will perform the exercise training three times per week, during 12 weeks, totaling 36 sections.

ELIGIBILITY:
Inclusion Criteria:

* Individuals resident in Porto Alegre and metropolitan area,
* aged ≥ 18 years;
* with diagnosis of heart failure class II and III (New York Heart Association);
* clinically stable at least 3 months prior to the start of the study;
* with left ventricular ejection fraction (LV) ≤ 45%;
* under optimized pharmacological treatment;
* with resting heart rate ˂ 120 bpm;
* resting blood pressure ˂ 180 / 110mm Hg;
* previously sedentary.

Exclusion Criteria:

* Decompensated heart failure (evidenced by ascites, lower limb edema, jugular swelling and / or pulmonary wheezing);
* individuals with decompensated metabolic diseases;
* acute coronary syndrome (ACS);
* survivors of sudden death;
* with acute myocardial infarction (AMI) and / or cardiac surgery for less than 6 months; -
* severe valvulopathies and / or cardiac arrhythmias;
* presence of asymmetric septal hypertrophic cardiomyopathy with dynamic outlet obstruction;
* with general contraindication criteria for performing the cardiopulmonary exercise test; -
* musculoskeletal disorders that limit exercise performance;
* with cognitive alterations that compromise the understanding of the stages and the execution of the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Capacity | After 12 weeks of training.
  Cardiopulmonary capacity assessed by peak oxygen consumption in treadmill cardiopulmonary exercise test.
Quality of life | After 12 weeks of training.
  Quality of life assessed by the Minnesota Living With Heart Failure Questionnaire. It is composed of 21 questions about limitations that are often associated with how heart failure interferes with patients' quality of life. The patient should consider the last month to answer the questions. The scale of responses for each question varies from 0 (zero) to 5, where 0 represents without limitations and 5, maximum limitation. These questions involve a physical dimension (from 1 to 7, 12 and 13 questions) that are highly interrelated with dyspnea and fatigue, an emotional dimension (17 to 21 questions) and other issues (8, 9, 10, 11, 14, 15 and 16 questions) which, added to the previous dimensions, form the total score. The scale totals 105 points. Higher values indicate maximum limitation and poorer quality of life.

SECONDARY OUTCOMES:
Functionality | After 12 weeks of training.
  Functionality assessed by the Duke Activity Status Index
Gait Speed | After 12 weeks of training.
  Gait Speed assessed by the Gait Speed Test.
Palmar Grip Strength | After 12 weeks of training.
  Palmar grip strength evaluated by dynamometry.
Maximum Inspiratory Pressure | After 12 weeks of training.
  Maximum inspiratory pressure evaluated by manovacuometry.
Endothelial Function | After 12 weeks of training.
  Endothelial function evaluated by brachial artery ultrasonography.
Lean Body Mass | After 12 weeks of training.
  Lean body mass assessed by arm muscle circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schaan, PhD, Principal Investigator — HCPorto Alegre
Locations (1):
- HCPortoAlegre, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] do Nascimento DM, Machado KC, Bock PM, Saffi MAL, Goldraich LA, Silveira AD, Clausell N, Schaan BD. Functional training improves peak oxygen consumption and quality of life of individuals with heart failure: a randomized clinical trial. BMC Cardiovasc Disord. 2023 Jul 29;23(1):381. doi: 10.1186/s12872-023-03404-7. PMID 37516830
- [Derived] do Nascimento DM, Machado KC, Bock PM, Saffi MAL, Goldraich LA, Silveira AD, Clausell N, Schaan BD. Cardiopulmonary exercise capacity and quality of life of patients with heart failure undergoing a functional training program: study protocol for a randomized clinical trial. BMC Cardiovasc Disord. 2020 Apr 25;20(1):200. doi: 10.1186/s12872-020-01481-6. PMID 32334527